CLINICAL TRIAL: NCT07072468
Title: A Randomized, Double-blind, Placebo-controlled Crossover Study to Evaluate Analgesic Efficacy, Safety and Tolerability of Repeated Doses of Topical VMD-3866 in Patients With Chemotherapy-induced Peripheral Neuropathy (CIPN)
Brief Title: Analgesic Efficacy and Safety of Topical VMD-3866 Gel in Management of Pain Induced by Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VM Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMT-03C; 119106 (Registry Identifier: IND Number; FDA, USA); 1011031 (Other: IRAS Number; Health Research Authority (HRA), UK)
Record Dates: First submitted 2025-05-30; First posted 2025-07-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Drug-Induced Nephropathy
Keywords: Chemotherapy-Induced Peripheral Neuropathy; Chemotherapy-Induced Peripheral Neuropathic Pain; Neuropathic Pain; Chronic Pain; Nephropathy; Tingling; Numbness; Burning; Drug-Induced Nephropathy
MeSH Terms: conditions — Neuralgia; Chronic Pain; Kidney Diseases; Paresthesia; Hypesthesia

STUDY DESIGN:
Intervention Model Description: Up to 16 participants is planned. Each participant will have 2 treatment periods, separated by a washout of at least 7 days. Participants will be randomized 1:1 to receive VMD-3866 gel in one period, and placebo gel in the other. Before the start of each treatment period, participants will have a Run-in period lasting 7 days, during which they will record numeric pain rating scale (NPRS) scores each morning in a trial diary. Participants will continue to record NPRS scores in the trial diary during treatment periods 1 and 2 (about 1 h after each dose).
  Eligible participants may attend an outpatient visit up to 14 days before their first dose of VMD-3866 or placebo, for baseline QST (quantitative sensory test) and, in ≥ 8 participants, a skin biopsy. Participants will visit the site for their first and last doses (Days 1 and 8) in each treatment period. All other doses they will self-administer at home. At the end of each treatment period, participants will undergo QST assessment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- VMD-3866 Gel (Experimental): Treatment Group
  Interventions: Drug: VMD-3866 Gel
- Placebo Gel (Placebo Comparator): Placebo Group
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: VMD-3866 Gel — Each participant will have 2 treatment periods, separated by a washout of at least 7 days. Participants will be randomized 1:1 to receive VMD-3866 gel in one period, and placebo gel in the other. Before the start of each treatment period, participants will have a Run-in period lasting 7 days, during which they will record NPRS scores each morning in a trial diary. Participants will continue to record NPRS scores in the trial diary during treatment periods 1 and 2 (about 1 h after each dose).
  Participants will be screened within 45 days before their first treatment period. Eligible participants may attend an outpatient visit up to 14 days before their first dose of VMD-3866 or placebo, for baseline QST and, in ≥ 8 participants, a skin biopsy. Participants will visit the site for their first and last doses (Days 1 and 8) in each treatment period. All other doses they will self-administer at home.
  Arms: VMD-3866 Gel
Drug: Placebo Gel — Each participant will have 2 treatment periods, separated by a washout of at least 7 days. Participants will be randomized 1:1 to receive VMD-3866 gel in one period, and placebo gel in the other. Before the start of each treatment period, participants will have a Run-in period lasting 7 days, during which they will record NPRS scores each morning in a trial diary. Participants will continue to record NPRS scores in the trial diary during treatment periods 1 and 2 (about 1 h after each dose). Participants will be screened within 45 days before their first treatment period. Eligible participants may attend an outpatient visit up to 14 days before their first dose of VMD-3866 or placebo, for baseline QST and, in ≥ 8 participants, a skin biopsy. Participants will visit the site for their first and last doses (Days 1 and 8) in each treatment period. All other doses they will self-administer at home.
  Arms: Placebo Gel

SUMMARY:
Peripheral neuropathy is a disorder caused by damage to the peripheral nerves. Chemotherapy-induced peripheral neuropathy (CIPN) is a common side effect of certain chemotherapy drugs, such as platinum-based compounds, taxanes, and vinca alkaloids, which can damage nerve fibres by disrupting their structure and function.

At present, relief of neuropathic pain in CIPN is limited, and existing therapies providing only modest and variable efficacy across patients.

This is a study of VMD-3866 gel (the study medicine), an experimental new topical medicine for treating pain caused by CIPN. The goal of this study is to assess if the study medicine improves pain symptoms in patients with CIPN, and to find out the side effects of the study medicine if any.

The study medicine will work by blocking certain proteins (called calcium channels) in the nerves under the skin which will lower the activity of the nerves and therefore reduce pain. Researchers will compare study medicine to a matching placebo (a look-alike gel that contains no drug) to see if VMD-3866 gel works to management of pain caused by CIPN.

DETAILED DESCRIPTION:
This is a Phase 2a double-blind, randomized, crossover repeated-dose trial of VMD-3866 topical gel in patients diagnosed with CIPN. Enrolment of up to 16 participants is planned.

Each participant will have 2 treatment periods, separated by a washout of at least 7 days. Participants will be randomized 1:1 to receive VMD-3866 gel in one period, and placebo gel in the other. Before the start of each treatment period, participants will have a Run-in period lasting 7 days, during which they will record NPRS scores each morning in a trial diary. Participants will continue to record NPRS scores in the trial diary during treatment periods 1 and 2 (about 1 h after each dose).

Participants will be screened within 45 days before their first treatment period. Eligible participants may attend an outpatient visit up to 14 days before their first dose of VMD-3866 or placebo, for baseline QST and, in ≥ 8 participants, a skin biopsy. Participants will visit the site for their first and last doses (Days 1 and 8) in each treatment period. All other doses they will self-administer at home. At the end of each treatment period, participants will undergo QST assessment and a skin biopsy if they had one at baseline. They will have a follow-up via telephone call 7-14 days after their last topical dose, or 7-14 days after the last skin biopsy (whichever is later).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient who has received any type of chemotherapy treatment for cancer and are in remission.

   Participants must be diagnosed with CIPN and must be showing moderate (Grade 2, as defined by the Common Terminology Criteria for Adverse Events) symptoms of peripheral sensory neuropathy, including pain and hypersensitivity, for ≥ 3 months. Participants must have had stable symptoms of CIPN for 8 weeks before screening. Participants with any other conditions associated with neuropathy, or conditions which might confound pain assessment (e.g. other severe pain or a skin condition in the area affected by neuropathy) will be excluded.
2. Aged 18-80 years (inclusive) at the time of consent.
3. Mean daily pain score of 4-8 on the 11-point NPRS, for at least 4 days during Run-in 1.
4. A score of 0 or 1 on the ECOG Performance Status Scale.
5. Capable of self-administering topical VMD-3866 or placebo gel to the designated treatment area(s).
6. Capable of understanding the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
7. Agrees to take only the allowed rescue medication (paracetamol) for breakthrough pain, from screening and throughout the study.
8. Willing to give written consent to participate after reading the informed consent form, and after having the opportunity to discuss the trial with the investigator or their delegate.
9. Agrees to follow the contraception requirements of the trial.
10. Agrees not to donate blood or blood products during the trial and for up to 3 months after the administration of the trial medication.

Exclusion Criteria:

1. Woman who is pregnant or lactating, or premenopausal woman who is sexually active and not using a reliable method of contraception.
2. History of painful conditions not associated with CIPN (e.g. frequent headache) that require administration of paracetamol or non-steroidal anti-inflammatory drugs, more than twice a week.
3. Presence of peripheral neuropathy of another etiology (e.g. alcohol, diabetes, toxins, neurotoxic treatments, hereditary, autoimmune).
4. Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the participant.
5. Clinical, history or previous laboratory evidence of significant conditions (e.g. diabetes, seizure or psychological conditions) that could interfere with completion of study procedures and assessments or pose an additional risk to the participant.
6. Cardiovascular events (stroke, heart attack, pulmonary embolism) in the last 3 months.
7. Significant psychiatric or neuropsychiatric disorders including but not limited to severe depression, dementia, bipolar disorder or schizophrenia spectrum disorder.
8. History of suicide attempt, or suicidal ideation in the last 6 months.
9. Presence of active and/or systemic infection, or history of severe infection during the 30 days prior to screening.
10. Damaged or tattooed skin, active skin disease, infection, severe erythema, or any other compromise in integrity of skin at the designated treatment area(s), which could influence or interfere with the evaluation of the safety or efficacy of VMD-3866.
11. Presence or history of severe adverse reaction(s) to any drug or a history of sensitivity to any excipients of VMD-3866.
12. Participation in any studies for skin irritation or sensitization within the 30 days before first dose.
13. If a skin biopsy is required: contraindications to skin biopsy (e.g. patients with significant bleeding tendencies or using anti-coagulants).
14. Receipt of an investigational medicinal product (including prescription medicines and devices) as part of another clinical trial, in the 3 months before first dose or 5-half-lives (whichever is longer); or is in the follow-up period of another clinical trial at the time of screening for this trial.
15. Use of topical capsaicin preparations (including Qutenza patch) in the 3 months before screening.
16. Use of opiate medication within the 28 days before screening.
17. Use of any pain medication (except the approved pain medications, see below), from 14 days before Run-in 1 to the last on-site study visit.

    Non-approved medications include; salicylates, NSAIDs, topical analgesic-containing gels or creams or patches, local treatment with anesthetics (such as lidocaine), steroids, or transcutaneous electric nerve stimulation.

    Approved medications include:
    * medications for the treatment of CIPN; gabapentin, pregabalin, amitriptyline, duloxetine, or a combination of those. The same medication/combination and dose should be used from 14 days before Run-in 1, until the end of the trial.
    * paracetamol can be used as a rescue medication for pain as required.
    * local anesthetic can be used prior to skin biopsy
18. Scheduled to undergo radiation therapy or cancer chemotherapy during the trial.

    Diagnostic/screening assessments
19. Blood pressure and pulse rate in supine position at the screening examination outside the following ranges: blood pressure 90-160 mm Hg systolic, 40-100 mm Hg diastolic; pulse rate 40_100 beats/min. If the values are out of range, one repeat is permitted. Patients can be included if the repeat value is within range.
20. QTcF > 450 msec (men) or > 470 msec (women) at Screening and pre-dose on Day 1. If the values are out of range, one repeat is permitted. Patients can be included if the repeat value is within range.
21. Positive test for hepatitis B, hepatitis C or HIV.

    Other
22. Presence or history of drug or alcohol abuse within the last 10 years, intake of > 14 units of alcohol weekly, smoking > 10 cigarettes daily, or heavy use of e-cigarettes (including vapes).
23. Evidence of drug abuse on urine testing.
24. Completion of <5 days in the 7-day Run-in 1 trial diary.
25. Objection by GP, on medical grounds, to patient entering trial.
26. Possibility that the patient will not cooperate with the requirements of the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the sum of daily numeric pain rating scale (NPRS) score at the end of each treatment period. | Daily for 8 days for each of 2 treatment periods, up to 1 month in total
  The participants assessed their current pain using the 11-point NPRS where: 0=no pain to 10=worst pain imaginable.
Number of participants with an Adverse Event (AE). | Daily for 8 days for each of 2 treatment periods, up to 1 month in total
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with AE(s) in each period will be reported.

SECONDARY OUTCOMES:
Change from baseline in average daily NPRS score, and the proportion of participants with at least 30% and 50% reductions | Daily for 8 days for each of 2 treatment periods, up to 1 month in total
  The participants assessed their current pain using the 11-point NPRS where: 0=no pain to 10=worst pain imaginable.
Change from baseline in the short-form McGill Pain Questionnaire 2 (SF-MPQ-2) | Day 1 and Day 8 for each of 2 treatment periods, up to 1 month in total
  The Short-form McGill Pain Questionnaire 2 (SF-MPQ-2) is a revised and expanded version of the original SF-MPQ, used to assess pain intensity and quality. It includes 22 descriptors of pain, with 11 sensory, 4 affective, and 7 neuropathic descriptors, rated on an 11-point numerical scale.
Change from baseline in weekly sleep interference scores assessed with Pain and Sleep Questionnaire three-item index (PSQ-3) | Day 1 and Day 8 for each of 2 treatment periods, up to 1 month in total
  The Pain and Sleep Questionnaire (PSQ-3) is a concise tool designed to evaluate the influence of pain on sleep quality. Each of the 3 items is scored individually on a 100 mm Visual Analog Scale (VAS), ranging from 0 (representing 'never') to 100 (indicating 'always'). The total score is obtained by summing up the scores of all three items, providing a comprehensive measure of the impact of pain on sleep quality. By quantifying the frequency of sleep disturbances attributed to pain, the PSQ-3 provides valuable insights into the intricate relationship between pain and sleep, crucial for assessing the holistic impact of myofascial low back pain on patients' well-being.
Patient global impression of change (PGIC) | Day 8 for each of 2 treatment periods, up to 1 month in total
  The PGIC is a scale participants use to rate the level of change they have experienced following treatment. The PGIC is a 7-point scale from 1 (very much better) to 7 (very much worse).
Frequency of use and dose of rescue medication during treatment period | Daily for each of 2 treatment periods, up to 1 month in total
  Number of days a participant used the rescue medication during the treatment period.
Reduction in cutaneous hypersensitivity as measured by the quantitative sensory test (QST) | Baseline on Day 1, and postdose on Day 8 of each of 2 treatment periods, up to 1 month in total
  QST is a non-invasive diagnostic method used to assess the level at which a subject reports sensing a physical stimulus (detection threshold) applied to the skin. It is measured using specific testing equipment and protocol, and the exact scoring can vary based on the specific equipment and protocol used. In general, lower thresholds (i.e., the patient detects the stimulus at lower intensities) may indicate heightened sensitivity, while higher thresholds may indicate reduced sensitivity. Changes in these thresholds over time can indicate a worsening of sensory dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Chair — VM Therapeutics LLC
Locations (1):
- Hammersmith Medicines Research Ltd (HMR code 24-503), London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HMR code 24-503; Safety and effectiveness of VMD-3866 in patients with CIPN (Protocol number VMT-03C) — http://www.hmrlondon.com